CLINICAL TRIAL: NCT01658982
Title: Cardiopulmonary Exercise Testing in Cirrhotic Patients: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, Assocaite Professor of Medicine, Mayo Clinic
Other Study IDs: 12-004215
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cirrhotic patients: cardiopulmonary exercise testing
  Interventions: Other: cardiopulmonary exercise testing

INTERVENTIONS:
Other: cardiopulmonary exercise testing — 3 minute step test compared to 6 minute bicycle test

SUMMARY:
Optimizing patient survival and organ utility is a constant struggle for the liver transplant community. Despite rigorous cardiovascular evaluation before liver transplantation cardiovascular events are one of the leading causes of post-transplant morbidity and mortality in both early and late post transplant periods. Poor performance on measures of cardiopulmonary fitness has been associated with worse outcomes in liver transplant candidates. The investigators seek to determine the feasibility of obtaining measures of cardiopulmonary performance in liver transplant candidates from standard cardiopulmonary exercise testing (CPET) and from a modified 3 minute step test and to determine whether the 3 minute step test is suitable for the assessment of cardiopulmonary fitness in a future outcome study.

DETAILED DESCRIPTION:
Subjects: 10 patients ≥40 years of age with cirrhotic end-stage liver disease undergoing liver transplantation evaluation at Mayo Clinic, Rochester, MN. Patients who require multi-organ transplant, or who have non-cirrhotic liver disease (neuroendocrine, amyloidosis, etc.) will be excluded. Each subject will undergo both standard CPET and modified 3 minute step test.

Exercise testing. Subjects will perform both tests during one visit to the cardiopulmonary research lab. A 30-60 minute period between tests will given. 5 patients will perform submaximal stress testing first and 5 will perform the full CPET first.

CPET: Patients will perform a 6 minute cardiopulmonary exercise test using the recumbent stationary bicycle facilitated by the co-investigators at the St Mary's cardiopulmonary exercise laboratory. Standard 12-lead electrocardiograms will be obtained at rest, each minute during exercise, and for at least five minutes during the recovery phase; blood pressure will be measured using a standard cuff sphygmomanometer. Minute ventilation (VE), breathing frequency (fR), tidal volume (VT), oxygen consumption (VO2), CO2 production (VCO2), RER, and end-tidal CO2 (PETCO2) will be obtained breath-by-breath and averaged over a 30-second period at rest and the last 30 seconds of each minute during exercise. In addition, heart rate (HR) and oxygen saturation (SaO2) will be obtained continuously using pulse oximetry. From these data, derived variables such as the VE/VCO2 ratio, oxygen pulse (VO2/HR) and an index of pulmonary capacitance (O2 pulse /[1/PETCO2]) are calculated at rest and during exercise. Ventilatory efficiency slopes (VE/VCO2 slope) [VE liter/min _ m (VCO2, liter/min) _ b], where m _ VE/VCO2 slope, and oxygen uptake efficiency slopes (OUES) [VO2, liter/min _ m (log10VE) _ b], where m _ OUES, are calculated using all exercise data points via least squares linear regression.

Modified 3 minute step test: Each participant will perform a sub-maximal exercise test that consists of 2 minutes of resting baseline, 3 minutes of step exercise, and 1 minute of recovery. Breathing pattern, gas exchange (as described above), and heart rate will be monitored using a simplified gas analysis system (SHAPE Medical Systems, Inc, St. Paul, MN). Submaximal testing will be defined by respiratory exchange ratio (RER), and perceived exertion (RPE). An exercise RER of 0.9 and RPE of 12 to 13 on the Borg scale (range, 6 to 20) is considered to be a sub-maximal level. At the end of the first & second minute of step exercise, RER and RPE will be recorded and the step rate adjusted (a patient with a low RER (< 0.8) and RPE (< 8) would increase the step rate for the second minute, whereas a patient with a higher RER (> 0.85) and RPE (> 11) would maintain the same step rate). On completion of the 3-minute step exercise, recovery data will be collected for 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* listed for liver transplantation with end stage liver disease

Exclusion Criteria:

* patients listed for liver transplant without end stage liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pre liver transpalnt patietns with cirrhosis and end stage liver disease
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
respiratory exchange ratio | during test

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Watt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States